CLINICAL TRIAL: NCT00002942
Title: Randomized Phase III Trial of G-CSF Primed Autologous Bone Marrow Versus Peripheral Blood Progenitor Cells (PBPC) as Hematopoietic Support for High-Dose Cyclophosphamide, Thiotepa, and Carboplatin (CTCb) Therapy in Poor Prognosis Breast Cancer
Brief Title: Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065391; CCCWFU-95496; NCI-G97-1145
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral Blood Progenitor Cells (Active Comparator)
  Interventions: Procedure: peripheral blood stem cell transplantation
- Autologous Bone Marrow Collection (Experimental)
  Interventions: Procedure: autologous bone marrow transplantation

INTERVENTIONS:
Procedure: autologous bone marrow transplantation
  Arms: Autologous Bone Marrow Collection
Procedure: peripheral blood stem cell transplantation
  Arms: Peripheral Blood Progenitor Cells

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with autologous bone marrow transplantation or peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Randomized phase III trial to compare bone marrow transplantation with peripheral stem cell transplantation following carboplatin in treating patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare engraftment rates using G-CSF primed autologous bone marrow vs PBCP as hematopoietic support following high dose CTCb for patients with poor prognosis breast cancer. II. Compare the complications of these two methods of hematopoietic progenitor cell collections. III. Compare Stage IV patients with bone or bone marrow involvement (assigned to PBPC collections) with Stage IV patients randomized to PBPC collections relative to the number of leukaphereses needed to collect the required number of progenitor cells as well as assess engraftment rates between these two groups. IV. Assess the response to high dose CTCb in this group of patients.

OUTLINE: All patients will receive G-CSF priming therapy for 5 consecutive days. Patients will then be randomized into two treatment arms: Arm 1 consists of autologous PBPC collection Arm 2 consists of autologous bone marrow collection Within 2 weeks after progenitor cell collection, all patients will receive high dose CTCb therapy by continuous infusion for 5 days, followed by autologous hematopoietic progenitor cell infusion at least three days later. G-CSF will also be given after infusion until ANC count is over 5,000 or over 1,000 for 3 consecutive days.

PROJECTED ACCRUAL: 66 patients will be accrued at a rate of 24 per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed Stage IIIB and IV adenocarcinoma of the breast Stage II-IIIA adenocarcinoma of the breast with poor risk features (including poorly differentiated histology, high mitotic rate, hormone receptor negative, high S phase) with at least three involved axillary lymph nodes, estimated five year relapse free survival rate less than 50%, and does not qualify for higher priority protocol treatments No central nervous system involvement

PATIENT CHARACTERISTICS: Age: 18 to 60 Performance status: Karnofsky 80-100% Life expectancy: Greater than 2 months Hematopoietic: Platelet count greater than 75,000/mm3 Neutrophils greater than 1500/mm3 Hepatic: Serum bilirubin, alkaline phosphatase, and SGOT or SGPT less than 3 times upper limit of normal, unless due to disease Renal: Serum creatinine less than 1.5 times upper limit of normal Creatinine clearance at least 60 mL.min Cardiovascular: Ventricular ejection fraction at least 45% No uncontrolled or severe cardiovascular disease, including recent myocardial infarction, congestive heart failure, angina, life threatening arrhythmia, or hypertension Pulmonary: DLCO and spirometry at least 50% of predicted Other: Not HIV positive Not HBsAG positive Not pregnant Must have functioning central venous catheter No active infection No uncontrolled diabetes mellitus No other prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior hematopoietic progenitor cell support Chemotherapy: No prior dose intensive therapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 1996-06; Primary Completion 2000-01 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David D. Hurd, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Acostamadiedo J, Case D, Perry J, et al.: Randomized trial of G-CSF primed (G') autologous bone marrow (ABM) vs. G' peripheral blood stem cells (PBSC) as hematopoietic support after high-dose cyclophosphamide (C) thiotepa (T), and carboplatin (CB) (CTCB) in poor prognosis breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A215, 56a, 2000.